CLINICAL TRIAL: NCT02107157
Title: Clinical and Histological Evaluation of the Picosure 755nm Laser With Cap Array for Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-PICO-CAPHST-ET
Record Dates: First submitted 2014-03-31; First posted 2014-04-08 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Facial Rejuvenation
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm Alexandrite laser with cap array (Experimental)
  Interventions: Device: 755nm Laser with Cap Array

INTERVENTIONS:
Device: 755nm Laser with Cap Array

SUMMARY:
The purpose of this study is to assess treatment of facial rejuvenation using the standard hand piece and a Lens Array for the 755nm Alexandrite laser.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 65 years old
2. Is willing to consent to participate in the study.
3. Is willing to comply with all requirements of the study including biopsies, being photographed, following post treatment care and attending all treatment and follow up visits.

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject is hypersensitive to light exposure OR takes photo sensitized medication.
3. The subject has active or localized systemic infections.
4. The subject has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy {greater than 81 mg per day}).
5. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. The subject has used Accutane within 6 months prior to enrollment.
8. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. The subject has a history of keloids.
11. The subject has evidence of compromised wound healing.
12. The subject has a history of squamous cell carcinoma or melanoma.
13. The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
14. The subject has an allergy to lidocaine and epinephrine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Dermatology and Laser Surgery, Sacramento, California, United States

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400
- See also: This is an explanation of the Fitzpatrick Skin typing that is described in the baseline characteristics section. — https://pubmed.ncbi.nlm.nih.gov/31896400/

RESULTS

PARTICIPANT FLOW:
Groups:
- 755nm Alexandrite Laser With Cap Array- Acne: 755nm Laser with Cap Array
  Treatment of acne in the facial region.
- 755nm Alexandrite Laser With Cap Array- Photodamage: 755nm Laser with Cap Array
  Treatment of photodamage in the facial region.
- 755nm Alexandrite Laser With Cap Array- Biopsy: 755nm Laser with Cap Array
  Biopsy samples were taken of subjects.
Period: Overall Study
Arm/Group | 755nm Alexandrite Laser With Cap Array- Acne | 755nm Alexandrite Laser With Cap Array- Photodamage | 755nm Alexandrite Laser With Cap Array- Biopsy
Started | 11 | 12 | 4
Completed | 6 | 11 | 4
Not Completed | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 755nm Alexandrite Laser With Cap Array- Acne; 755nm Alexandrite Laser With Cap Array- Photodamage; 755nm Laser With Cap Array- Biopsy: 755nm Laser with Cap Array
- Total: Total of all reporting groups
Arm/Group | 755nm Alexandrite Laser With Cap Array- Acne | 755nm Alexandrite Laser With Cap Array- Photodamage | 755nm Laser With Cap Array- Biopsy | Total
Number analyzed (Participants) | 10 | 12 | 4 | 26
Age, Categorical [Count of Participants; unit: Participants] — Population: One subject in the acne group withdrew from the study before the first treatment occurred and baseline information was collected. The withdrawal was due to scheduling conflicts.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 10 | 12 | 3 | 25
    >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject in the acne group withdrew from the study before the first treatment occurred and baseline information was collected. The withdrawal was due to scheduling conflicts.
  Participants
    Female | 10 | 12 | 1 | 23
    Male | 0 | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One subject in the acne group withdrew from the study before the first treatment occurred and baseline information was collected. The withdrawal was due to scheduling conflicts.
  Participants
    Race/Ethnicity: Caucasian | 4 | 9 | 3 | 16
    Race/Ethnicity: Hispanic | 4 | 1 | 0 | 5
    Race/Ethnicity: Asian | 2 | 2 | 1 | 5
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is. Population: One subject in the acne group withdrew from the study before the first treatment occurred and baseline information was collected. The withdrawal was due to scheduling conflicts. Additionally, one subject in the acne group did not fill out Fitzpatrick Skin Type. The subject missing this baseline information withdrew from the study before the first treatment occurred due to scheduling conflicts.
  Participants
    number analyzed (Participants) | 9 | 12 | 4 | 25
    Fitzpatrick Skin Type I | 0 | 0 | 0 | 0
    Fitzpatrick Skin Type II | 2 | 0 | 2 | 4
    Fitzpatrick Skin Type III | 4 | 8 | 1 | 13
    Fitzpatrick Skin Type IV | 3 | 4 | 1 | 8
    Fitzpatrick Skin Type V | 0 | 0 | 0 | 0
    Fitzpatrick Skin Type VI | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Facial Scarring Score
Description: Physicians will examine the subjects' facial scarring using the Physician Global Scarring Grading (PGSG) scale. This scale counts and types scars by tallying up of the number and severity of the scars according to an organized grading system, where 0 is the lowest point value and represents no scarring. The theoretical highest score possible is an 84. The change in the score from the baseline to the follow up was collected. A negative change indicates a decrease in points (which indicates improvement).
Time Frame: Baseline and 3 months post last treatment
Population: 4 subjects withdrew due to scheduling conflicts, and 1 moved out of state. 1 subject had completed the photoaging scoring sheet instead of the acne scarring scoring sheet for their followup, so their scores are not reported. 1 subject is missing data, so their score cannot be used.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser With Cap Array- Acne
Number analyzed (Participants) | 4
score on a scale | -.50 (1)

2. Primary Outcome: Photodamage Score Change
Description: The photodamage is assessed by examining fine wrinkles, mottled hyperpigmentation, and overall integrated assessment of photodamage. These 3 categories are broken down into their own scales of 0 to 4 based on severity. 0 indicates none, 1 indicates minimal, 2 indicates mild, 3 indicates moderate, and 4 indicates severe. The total points from all 3 categories added up will range from 0 to 12, where 12 is the most photodamage possible. A decrease in score indicates less photodamage.
Time Frame: Baseline and 3 months post last treatment
Population: 1 subject withdrew from the study due to scheduling conflicts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser With Cap Array- Photodamage
Number analyzed (Participants) | 11
score on a scale | -.363 (1.20)

3. Primary Outcome: Number of Participants With Signs of New Collagen Generations
Description: Subjects will have one 3mm punch biopsy obtained pretreatment from an inconspicuous area and subsequent biopsies at one or any of the following visits after treatment. Pathologies will be provided by pathologists who are able to determine any developments of dermal mucus, dermal elastic fibers, or changes in collagen III. An increase in any of these categories corresponds with skin rejuvenation.
Time Frame: 3 months post last treatment
Population: 2 other patients had biopsies performed on them, but did not come in for a biopsy follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | 755nm Alexandrite Laser With Cap Array- Biopsy
Number analyzed (Participants) | 2
Participants
  dermal mucus increased | 2
  dermal elastic fibers increased | 2
  collagen III increased | 2

ADVERSE EVENTS:
Time Frame: Adverse Events occurring will be captured and followed for study duration, approximately 13 months.
Groups:
- 755nm Alexandrite Laser With Cap Array- Biopsy: 755nm Laser with Cap Array
Arm/Group | 755nm Alexandrite Laser With Cap Array- Acne | 755nm Alexandrite Laser With Cap Array- Photodamage | 755nm Alexandrite Laser With Cap Array- Biopsy
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 8/11 | 12/12 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 755nm Alexandrite Laser With Cap Array- Acne (N=11) | 755nm Alexandrite Laser With Cap Array- Photodamage (N=12) | 755nm Alexandrite Laser With Cap Array- Biopsy (N=4)
redness (Skin and subcutaneous tissue disorders) | 8 | 12 | 0
edema (Skin and subcutaneous tissue disorders) | 8 | 12 | 0
Pinpoint Bleeding (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acne breakout (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.